CLINICAL TRIAL: NCT03086941
Title: The Use of Supraglottic I-Gel Airway as a Conduit for Fiberoptic Guided and Blind Intubation in Children
Brief Title: Blind Versus Fiberoptic Intubation Through I-GEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Galal EL-Sherbeny, Assistant lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: N-60-2016
Record Dates: First submitted 2017-03-11; First posted 2017-03-22 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: I-gel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B(blibd) (Active Comparator): group B (blind); an appropriate size endotracheal tube will be introduced through I-gel blindly. Only smooth intubation without force together with manoeuvres necessary to correct the position of tracheal tube will be allowed. Only one attempt of blind intubation is allowed to avoid airway injury. Any resistance to first attempt tube insertion will indicate failure of blind tube insertion.
  Interventions: Device: I-gel
- Group C(control) (Active Comparator): group C (control), a paediatric fibrescope will be primed with an appropriate size tracheal tube. The fibrescope will be introduced through I-gel and guide tracheal intubation. After insertion of tube and confirmation of position, the fiberscope will be removed
  Interventions: Device: I-gel

INTERVENTIONS:
Device: I-gel — To compare between use of I-gel as a conduit for blind intubation and as a conduit for fiberoptic guided intubation in children. We also aim to validate the use of I-gel as conduit for blind intubation in absence of fiberoptic or lack of experience of its use.

SUMMARY:
Aim of the work

To compare between use of I-gel as a conduit for blind intubation and as a conduit for fiberoptic guided intubation in children and also aim to validate the use of I-gel as conduit for blind intubation in absence of fiberoptic or lack of experience of its use.

Objectives:

* To validate I-gel use as blind intubating conduit in children.
* To Estimate the duration of blind intubation using I-gel and duration of fiberoptic guided intubation through I-gel.

Ethical Considerations

The study protocol will be approved by the Research Ethics Committee.

DETAILED DESCRIPTION:
Introduction:

A supraglottic airway device is designed to maintain a clear airway while sitting above, and creating a seal around the larynx. It may be used in elective surgery, as an airway rescue device in failed tracheal intubation, as a conduit for tracheal intubation, or in emergencies such as cardiorespiratory arrest, both in and out of hospital.

'First-generation'supraglottic airway devices are simple airway tubes such as the laryngeal mask airway (LMA) Classic. 'Second generation' devices contain suction ports and integral bite blocks, these include the LMA Proseal and the i-gel.

The I-gel is the innovate second generation supraglottic airway and it is considered the first major development since LMA. The I-gel has changed the face of airway management and is now widely used in anesthesia and resuscitation across the globe. It is made from a medical grade thermoplastic elastomer and it is designed to create a non-inflatable, anatomical seal of the pharyngeal, laryngeal and perilaryngeal structures.

Pediatrics are not small adults, there are a number of anatomical differences which make airway management difficult than adults. Predicatably, these differences are most pronounced at birth and the most unfamiliar(non-adult like) airway is encountered in neonates and infants under 1 year of age.

Aim of the work

To compare between use of I-gel as a conduit for blind intubation and as a conduit for fiberoptic guided intubation in children and also aim to validate the use of I-gel as conduit for blind intubation in absence of fiberoptic or lack of experience of its use.

Objectives:

* To validate I-gel use as blind intubating conduit in children.
* To Estimate the duration of blind intubation using I-gel and duration of fiberoptic guided intubation through I-gel.

Ethical Considerations

The study protocol will be approved by the Research Ethics Committee.

Methodology

I. Study design

Prospective randomized controlled trial (non inferiority design)

II. Study setting and location

The study will be conducted in Children Hospital of Cairo University.

III. Study population

This Study will be conducted on 88 children aged from one to ten years presented for elective surgical procedure at Children Hospital of Cairo University. Patient will be divided into two equal groups; group C control group (n=44) and group B (blind) (n=44).

V. Study Procedures

1. Randomization (in RCT only) Once enrolled in the study, patients will be randomly assigned into two groups; fiberoptic guided (control) group (Group C: n= 44), blind group (Group B: n=44). Randomization will be done using computer generated number and concealed using sequentially numbered, sealed opaque envelope.
2. Study Protocol Randomization will be done by computer generated numbers and concealed by serially numbered, opague and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. Prior to surgery the appropriate numbered envelopes will be opened by the nurse, the card inside will determine the patient group.

   All children will be premedicated with oral midazolam 0.5mg/kg Half hour before procedure and atropine at a dose of 0.02mg/kg (IM). Continuous electrocardiogram (ECG), pulse oximetry, non-invasive arterial blood pressure, and temperature monitoring will be applied and all patients will be induced with inhalational anesthetic using Sevoflurane + oxygen (O2) and I.V line will be inserted. After deepening of the anesthesia, fentanyl 1μg/kg, and muscle relaxant will be given in the form of atracurium 0.5mg/kg.

   The absence of mydriasis, divergent gaze, haemodynamic or motor response to the jaw thrust manoeuvre will be used as parameters to guide adequate depth of anesthesia(7). Supraglottic I-gel of appropriate size (according to body wight) will be inserted after lubrication with K-Y Lubricating Jelly (Johnson & Johnson Medical Limited, Gargrave, Skipton, UK). Air way manoeuvres like jaw thrust or head tilt will be used to facilitate insertion.

   Adequate ventilation will be confirmed by adequate chest expansion and capnography waveform. If ventilation is adequate, the SG I-gel will be secured. In case of inadequate ventilation after I-gel insertion, airway manoeuvres like adjusting head/neck position and changing depth of insertion can be used to improve ventilation.A maximum of three SGA insertion attempts will be allowed then conventional laryngoscopic intubation will be performed.

   After securing SG I-gel, according to patients group; in group C (control), a paediatric fibrescope will be primed with an appropriate size tracheal tube. The fibrescope will be introduced through I-gel and guide tracheal intubation. After insertion of tube and confirmation of position, the fiberscope will be removed

   In group B (blind); an appropriate size endotracheal tube will be introduced through I-gel blindly. Only smooth intubation without force together with manoeuvres necessary to correct the position of tracheal tube will be allowed. Only one attempt of blind intubation is allowed to avoid airway injury. Any resistance to first attempt tube insertion will indicate failure of blind tube insertion.

   In both groups, a second person will stabilise the SG I-gel in the set position in order to prevent unintentional movement during the intubation procedure and removal of I-gel. Tube insertion will be confirmed by capnography, fibrescope and bilateral air entry by auscultation after connection of breathing circuit. To remove the SG I-gel after successful intubation, the breathing circuit will be disconnected, and the I-gel will be withdrawn with the aid of a stylet (stabilizer) in a continuous push-pull movement. If saturation fall below 92%, or if facemask ventilation or ventilation via the SGA begin to fail, this indicate securing airway with conventional intubation
3. Measurement tools

   * Patients demographic data will be collected; age, gender, weight, height and type of surgery.
   * The success rate and number of attempts of SG I-gel insertion will be recorded and the time taken for insertion from removal of face mask until appearance of end-tidal CO2 on the monitor after connection of the breathing circuit to the SG I-gel.
   * The success rate of first attempt intubation and time taken for tube insertion from start of tube introduction till appearance of appearance of end-tidal CO2 on the monitor after connection of the breathing circuit to the tube will be recorded.
   * Adverse events will be recorded ; suspicion of aspiration or regurgitation, hypoxia, bronchospasm, laryngospasm and coughing. Staining of blood on the SG I-gel will be recorded, as well as dental, tongue or lip trauma.
   * Postoperative dysphagia, sore throat and hoarseness of voice will be recorded.

VI. Study outcomes

1. Primary outcome

   * The success rate of first attempt intubation
2. Secondary outcome(s)

   * The success rate of SG I-gel insertion
   * Number of trials of I-gel insertion with maximum three trials.
   * Time taken for I-gel insertion.
   * Time taken for endotracheal tube insertion.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I-II
2. Age (2-6)

Exclusion Criteria:

1. Known difficulty of intubation. (Airway assessment clinically for presence of retrognathia, small mandibular cavity, limited neck or mandibular mobility and presence of syndromes associated with facial abnormalities e.g Pierre Robin sequence, Treacher Collins, Hurler's Hunter's syndrome (mucopolysaccharidoses), Beckwith-Wiedemann syndrome and Down's syndrome.)
2. Emergency surgery.
3. Risk of aspiration (e.g; full stomach, GERD, CHPS).
4. Respiratory tract infections.
5. Children not fitted with I-Gel.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
The success rate of first attempt intubation | The success rate for insertion will be recorded 5 minutes after induction of anesthesia
  assessing the success rate of first attempt to insert the endotracheal tube through I-gel either blindly or by a fiberscope

CONTACTS AND LOCATIONS:
Overall Officials: Amr Sherbeny, Master, Principal Investigator — Research Ethics Committee
Locations (1):
- Children Hospital of Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided